CLINICAL TRIAL: NCT02841683
Title: Evaluation of Effectiveness of Tabac Info Service (EE-TIS)
Brief Title: Pragmatic Randomised Controlled Trial Evaluating Effectiveness of a Smoking Cessation e- Intervention " Tabac Info Service "
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole des Hautes Etudes en Santé Publique (Other)
Responsible Party: Principal Investigator, Linda Cambon, Professor, Ecole des Hautes Etudes en Santé Publique
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cnamts_2016_1
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle counseling (Active Comparator): A smoking cessation E-intervention, Tabac Info Service (TIS), by website and mobile application
  Interventions: Behavioral: Tabac Info Service
- Current practices (No Intervention): Current practices of smoking cessation in France

INTERVENTIONS:
Behavioral: Tabac Info Service — A smoking cessation E-intervention, Tabac Info Service (TIS), by website and mobile application
  Arms: Lifestyle counseling

SUMMARY:
Introduction - A national smoking cessation E-intervention, called Tabac Info Service (TIS), was developed in France to provide an adapted web and mobile application support to smoking cessation for all adults smokers, with or without chronic diseases, who want to stop smoking. This paper presents the study protocol of the evaluation of the program. The primary objective of this evaluation is to assess the efficacy and efficacy conditions of eTIS. The secondary objectives are to 1) describe efficacy variations in regard to user characteristics, 2) analyze mechanisms and efficacy conditions of eTIS, through variations of use, social or environmental contextual factors likely to influence the efficacy of eTIS, and the behavior change techniques (BCTs).

Methods and analyses - The study design is a two-arm pragmatic randomized controlled trial including a process evaluation with at least 3000 participants randomized to the intervention or to the control arm (current practices presented in a non-interactive website). Inclusion criteria are: Adults, Smokers with an information and consent form completed, Getting a smartphone and using mobile applications, wanting stop to smoking in short, medium or long terms. The exclusion criterion is the refusal to participate in the study. The primary outcome is the point prevalence abstinence of 7 days at 6 months later. The secondary outcomes are: the point prevalence abstinence of 24 h at 3 months later, the point prevalence abstinence of 30 days at 12 months later, number of quit attempts during the study, progression of stages within the program (changes and duration in each stage). Data will be analyzed in Intention to treat (main analyze) and per protocol ways. A logistic regression will be carried out to estimate an OR [95% confidence interval] for efficacy. A multivariate multilevel analysis will explore the influence of patients' characteristics, social and environmental context, conditions of use and behavior change techniques on results.

Dissemination -The findings of this study will allow us to understand and characterize the efficacy of eTIS, and conditions of its efficacy, underlining psychological, sociological, environmental and contextual factors, which could influence the efficacy of this type of intervention on smokers. These findings will be disseminated through peer-reviewed journals, national and international conference presentations and public events.

ELIGIBILITY:
Inclusion Criteria:

* adult smokers
* with an information and consent form completed
* agreed to participate in the study
* get a Smartphone and be willing to use applications
* wanting stop smoking (in short, medium or long terms).

Exclusion Criteria:

* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2806 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence of 7 days | 6 months

SECONDARY OUTCOMES:
continuous abstinence rate | 6 months
  Defined as the proportion of participants remaining continuously abstinent from the cessation date to the endpoint
continuous abstinence rate | 12 months
  Defined as the proportion of participants remaining continuously abstinent from the cessation date to the endpoint
minimum 24-hour point abstinence | 3 months
minimum 30-day point abstinence | 12 months
number of quit attempts | 6 months
total duration of quit attempts | 6 months
  calculated as sum of days with no use

CONTACTS AND LOCATIONS:
Locations (1):
- université de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Affret A, Luc A, Baumann C, Bergman P, Le Faou AL, Pasquereau A, Arwidson P, Alla F, Cambon L. Effectiveness of the e-Tabac Info Service application for smoking cessation: a pragmatic randomised controlled trial. BMJ Open. 2020 Oct 27;10(10):e039515. doi: 10.1136/bmjopen-2020-039515. PMID 33109670
- [Derived] Cambon L, Bergman P, Le Faou A, Vincent I, Le Maitre B, Pasquereau A, Arwidson P, Thomas D, Alla F. Study protocol for a pragmatic randomised controlled trial evaluating efficacy of a smoking cessation e-'Tabac Info Service': ee-TIS trial. BMJ Open. 2017 Feb 24;7(2):e013604. doi: 10.1136/bmjopen-2016-013604. PMID 28237958